CLINICAL TRIAL: NCT02558361
Title: A Skin and Synovial Tissue Assessment of Overlapping Genes and Their Response After 3 Months Treatment With Apremilast in Patients With Psoriatic Arthritis
Brief Title: Treatment With Apremilast in Patients With Psoriatic Arthritis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: FDA approved synovial biopsy device unavailable
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00023672
Record Dates: First submitted 2015-09-16; First posted 2015-09-24 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-06

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Therapeutics; apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label, single arm (Other): Baseline visit:assess disease activity,synovial tissue biopsy of the knee with active synovitis [target joint] and punch skin biopsy of a target psoriatic plaque. Perform a similar punch skin biopsy on adjacent normal skin. Start apremilast (standard dosing). Perform venipuncture: blood samples will be obtained for routine studies, quantitative RT-PCR & ex vivo cytokine production assays. UA/pregnancy test.
  Month 1: assess disease active , monitor for AE's; repeat punch skin biopsy of target psoriatic plaque. Blood samples will be obtained for RT-PCR and ex vivo cytokine production assays.
  Month 3: same as month 1; repeat synovial tissue biopsy from target knee joint and punch skin biopsy on target psoriatic plaque. Blood samples for RT-PCR ex vivo cytokine production assays and routine studies.
  Interventions: Drug: Treatment with Apremilast

INTERVENTIONS:
Drug: Treatment with Apremilast — Standard dosing with apremilast (Otezla) will be used. [30mg po BID after initial titration]
  Other Names: Otezla

SUMMARY:
Apremilast (Otezla®) is a Federal Drug Administration (FDA)-approved treatment for psoriatic arthritis and psoriasis. Although there are a lot of data demonstrating how apremilast works in the laboratory, there are very few demonstrating how it works in the actual target organ, i.e. the skin or synovial (joint) tissue in patients with psoriasis and psoriatic arthritis.

Laboratory data has demonstrated that apremilast decreases inflammatory proteins and increases anti-inflammatory proteins. However, almost all of these data/studies have been performed on the blood of patients with psoriasis and psoriatic arthritis, not the skin or synovial (joint) tissue. These studies that have been performed on the blood of patients with this condition may, or may not, reflect the true response to therapy in the synovial (joint) tissue and/or skin.

DETAILED DESCRIPTION:
Purpose of the study Apremilast (Otezla®) is a Federal Drug Administration (FDA)-approved treatment for psoriatic arthritis and psoriasis. Although there are a lot of data demonstrating how apremilast works in the laboratory, there are very few demonstrating how it works in the actual target organ, i.e. the skin or synovial (joint) tissue in patients with psoriasis and psoriatic arthritis.

Laboratory data has demonstrated that apremilast decreases inflammatory proteins and increases anti-inflammatory proteins. However, almost all of these data/studies have been performed on the blood of patients with psoriasis and psoriatic arthritis, not the skin or synovial (joint) tissue. These studies that have been performed on the blood of patients with this condition may, or may not, reflect the true response to therapy in the synovial (joint) tissue and/or skin. They also provide no data regarding the timing of response in the target organs.

Because of these limitations in the existing literature, a study assessing the response to apremilast in synovial (joint) tissue and skin is needed. This will be a small study assessing the inflammatory response in the synovial (joint) tissue and skin samples from patients with psoriatic arthritis and psoriasis. These data will be very important in demonstrating the effect of apremilast on the target organ tissues; i.e. synovial (joint) tissue and skin.

We are asking you to take part in this research study because you have both psoriasis and psoriatic arthritis. Both conditions are active and you are an appropriate candidate to be treated with apremilast, i.e. this same treatment would be offered to you if you were not to enroll in this study. You are also an appropriate candidate to receive skin and synovial (joint) tissue biopsies. We want to find out how specific proteins in your skin and synovial (joint) tissue that are responsible for the inflammation associated with psoriasis and psoriatic arthritis respond to treatment with apremilast.

Study Procedures: What will happen during this study?

This study will consist of three study visits over a period of three months. If appropriate, you will be started on apremilast at your first study visit. This is part of your standard of care. The dose of apremilast you will receive will be the normal FDA-approved dose. You will not receive a placebo (sugar) pill. Everyone who participates in the study will be treated with apremilast. The study procedures that will take place at each of the three visits are listed below:

Baseline Visit:

Review inclusion/exclusion criteria Medical history obtained by the study nurse A physical examination by the study doctor Obtain blood and urine samples with psoriatic arthritis and psoriasis. These data will be very important in demonstrating the effect of apremilast on the target organ tissues; i.e. synovial (joint) tissue and skin.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Must be in general good health (except for psoriatic arthritis and psoriasis) as judged by the Investigator, based on medical history, physical examination, clinical laboratories, and urinalysis. (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions).
2. Patients at least 18 years of age with PsA (must meet CASPAR Criteria) and PsO.
3. Active knee synovitis (target joint)
4. Active psoriatic plaque (target skin lesion)
5. Not currently taking or previously on Otezla
6. Cannot be on concurrent biologics
7. Females of childbearing potential (FCBP)† must have a negative pregnancy test at Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive§ options described below:

Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]; PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (male latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]) while on investigational product and for at least 28 days after the last dose of investigational product.

† A female of childbearing potential is a sexually mature female who 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or 2) has not been postmenopausal for at least 24 consecutive months (that is, has had menses at any time during the preceding 24 consecutive months).

§ The female subject's chosen form of contraception must be effective by the time the female subject is randomized into the study (for example, hormonal contraception should be initiated at least 28 days before randomization).

Exclusion Criteria:

* The presence of any of the following will exclude a subject from enrollment:

  1. Other than psoriatic arthritis, any clinically significant (as determined by the Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled.
  2. Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study.
  3. Prior history of suicide attempt at any time in the subject's life time prior to screening or randomization, or major psychiatric illness requiring hospitalization within the last 3 years.
  4. Pregnant or breast feeding.
  5. Active substance abuse or a history of substance abuse within 6 months prior to Screening.
  6. Malignancy or history of malignancy, except for:

     treated [ie, cured] basal cell or squamous cell in situ skin carcinomas; treated [ie, cured] cervical intraepithelial neoplasia (CIN) or carcinoma in situ of cervix with no evidence of recurrence within the previous 5 years.
  7. Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half lives, if known (whichever is longer).
  8. Prior treatment with apremilast.
  9. Currently treated with a biologic (TNFi)
  10. Standard exclusions for treatment or biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Comparison of the change in the specific 32 gene products as measured by RT-PCR from baseline to Month 3 on synovial, skin samples (Co-primary endpoints) using the sign test. | To be assessed by a change from baseline to month three

SECONDARY OUTCOMES:
Comparison of the change in the RT-PCR gene products from baseline to Month 3 on blood samples (sign test). | To be assessed by a change from baseline to month three

OTHER OUTCOMES:
Comparison of the change in the RT-PCR gene products from baseline to month 1 on skin samples (sign test). | To be assessed by a change from baseline to month three
Comparison of the change in the RT-PCR gene products of lesional skin to normal skin at baseline (sign test). | To be assessed by a change from baseline to month three
Comparison of a change in all the markers of disease activity from baseline to month 3 (sign tests). | To be assessed by a change from baseline to month three

CONTACTS AND LOCATIONS:
Overall Officials: John D Carter, MD, Principal Investigator — University of South Florida Morsani College of Medicine
Locations (1):
- Morsani Center for Advanced healthcare, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No